CLINICAL TRIAL: NCT03941886
Title: Implementation of First-trimester Screening and Prevention of Preeclampsia: a Stepped Wedge Cluster-randomized Trial in Asia
Brief Title: Implementation of First-trimester Screening and preventiOn of pREeClAmpSia Trial (FORECAST)
Acronym: FORECAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiu Yee Liona Poon (Other)
Responsible Party: Sponsor-Investigator, Chiu Yee Liona Poon, Professor (Clinical), Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0434
Record Dates: First submitted 2018-12-19; First posted 2019-05-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia; Aspirin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster-randomized trial. There are total of 7 clusters across Asia. This study involves a period where no intervention will take place at all recruiting units, i.e. routine prenatal care, and then at regular intervals (every 6 weekly), one cluster will be randomized to transit from non-intervention group to intervention group in which first-trimester screening for preterm-preeclampsia by the Bayes based method followed by commencement of low-dose aspirin prophylaxis for high-risk women.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-intervention group (No Intervention): Participants receive routine prenatal care
- Intervention group (Experimental): Participants receive first-trimester screening for preterm-preeclampsia by the Bayes based method followed by commencement of low-dose aspirin prophylaxis in high-risk women.
  Interventions: Other: Low-dose aspirin in women with high risk of preeclampsia

INTERVENTIONS:
Other: Low-dose aspirin in women with high risk of preeclampsia — Low-dose aspirin 150-162 mg/night or 100 mg/night if body weight <40 Kg, from <15 weeks till 36 weeks or, in the event of early delivery, at the onset of labor
  Arms: Intervention group

SUMMARY:
This implementation study aims to evaluate the efficacy, acceptability, and safety of first-trimester screening and prevention for preterm-preeclampsia. It is a multicenter stepped wedge cluster randomized trial including maternity / diagnostic units from ten regions in Asia. The study involves a period where no intervention will take place at all recruiting units, and then at regular intervals, one cluster will be randomized to transit from non-intervention group to intervention group in which first-trimester screening for preterm-preeclampsia by the Bayes based method followed by the commencement of low-dose aspirin in high-risk women.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy;
* Live fetus;

Exclusion Criteria:

* Multiple pregnancy;
* Major fetal defects identified at 11-13 weeks of assessment;
* Non-viable fetus (missed spontaneous abortion or stillbirth).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42454 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Delivery with preterm-preeclampsia | Before 37 weeks of gestation
  Proportions of delivery with preterm preeclampsia between non-intervention and intervention groups

SECONDARY OUTCOMES:
Adverse outcomes with delivery at <34, <37 and ≥37 weeks of gestation | at <34, <37 and ≥37 weeks of gestation
  including preeclampsia, gestational hypertension, small for gestational age birth weight (<5th percentile), stillbirth, placental abruption
Neonatal mortality | during the first 28 days of life (0-27 days)
  A neonatal death is a death during 0-27 days of life. Composite neonatal morbidity (any one of the following): > grade II intraventricular hemorrhage; neonatal sepsis confirmed by cultures; neonatal anemia requiring transfusion; respiratory distress syndrome requiring surfactant and ventilation; necrotising enterocolitis requiring surgical intervention.
  Composite neonatal therapy (any one of the following): Neonatal high dependency or intensive care unit admission; Ventilation - need of positive pressure or intubation.
Low birth weight | at birth
  Low birth weight <3rd, 5th and 10th percentile
Stillbirth | at or after 20 to 28 weeks of pregnancy
  Fetal death at or after 20 to 28 weeks of pregnancy
Spontaneous preterm birth | At <34 and <37 weeks' gestation
  Spontaneous preterm birth (SPB) includes preterm labor, preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM) and cervical weakness; it does not include indicated preterm delivery for maternal or fetal conditions.
Acceptability for PE screening | in the first trimester of pregnancy (11-13 weeks of gestation)
  If subjects are under the intervention group upon proper consent procedure is done, at 11-13 weeks of gestation, the procedures below will be done.
  1. Collection of maternal information (obstetrical, medical and drug history including aspirin intake with indication)
  2. Measurement of maternal MAP and UtA-PI will be measured according to standardized protocols.
  3. Blood sample will be drawn to determine of serum level of PIGF.
  The individual study participant's risk of preterm-PE will be computed using the Bayes based method.
Acceptability for aspirin treatment. | from <15 weeks till 36 weeks of gestation or, in the event of early delivery, at the onset of labor
  When patients are subjected to be high risks in preeclampsia screening, they will be asked if they accept the aspirin for treatment. If they do not accept, they will continue with routine care. The willingness of subjects will all be recorded on the Case report forms for data collection.
Composite neonatal morbidity | during the first 28 days of life (0-27 days)
  Composite neonatal morbidity (any one of the following): > grade II intraventricular hemorrhage; neonatal sepsis confirmed by cultures; neonatal anemia requiring transfusion; respiratory distress syndrome requiring surfactant and ventilation; necrotising enterocolitis requiring surgical intervention.
Composite neonatal therapy | during the first 28 days of life (0-27 days)
  Composite neonatal therapy (any one of the following): Neonatal high dependency or intensive care unit admission; Ventilation - need of positive pressure or intubation.
Gestational age at delivery | at delivery
  Gestational age at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Liona CY Poon, MD, Principal Investigator — Chinese University of Hong Kong
Locations (19):
- China (3):
  - Guangzhou Women and Children's Medical Center, Guangzhou
  - Kunming Angel Women & Children Hospital, Kunming
  - Nanjing Drum Tower Hospital, Nanjing
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong, Hong Kong, China
  - Kwong Wah Hospital, Hong Kong
- Harapan Kita Hospital, Jakarta, Indonesia
- Japan (3):
  - Clinical Research Institute of Fetal Medicine, Osaka
  - Showa University Hospital, Tokyo
  - Japan Society for the Study of Hypertension in Pregnancy, Toyama
- Pusat Perubatan Universiti Kebangsaan Malaysia (UKM) Medical Centre, Bandar Tun Razak, Malaysia
- Philippine General Hospital, Manila, Philippines
- National University Hospital, Singapore, Singapore
- Taiwan (2):
  - Chang Gung Hospital, Taipei
  - Taiji Clinic, Taipei
- Thailand (4):
  - Chulalongkorn University Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Khlong Luang
- Hanoi Obstetrics & Gynecology Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geographic variation in the incidence of hypertension in pregnancy. World Health Organization International Collaborative Study of Hypertensive Disorders of Pregnancy. Am J Obstet Gynecol. 1988 Jan;158(1):80-3. PMID 2962500
- [Background] Steegers EA, von Dadelszen P, Duvekot JJ, Pijnenborg R. Pre-eclampsia. Lancet. 2010 Aug 21;376(9741):631-44. doi: 10.1016/S0140-6736(10)60279-6. Epub 2010 Jul 2. PMID 20598363
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Tranquilli AL, Dekker G, Magee L, Roberts J, Sibai BM, Steyn W, Zeeman GG, Brown MA. The classification, diagnosis and management of the hypertensive disorders of pregnancy: A revised statement from the ISSHP. Pregnancy Hypertens. 2014 Apr;4(2):97-104. doi: 10.1016/j.preghy.2014.02.001. Epub 2014 Feb 15. No abstract available. PMID 26104417
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Hypertension in Pregnancy: The Management of Hypertensive Disorders During Pregnancy. London: RCOG Press; 2010 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK62652/ PMID 22220321
- [Background] Committee Opinion No. 638: First-Trimester Risk Assessment for Early-Onset Preeclampsia. Obstet Gynecol. 2015 Sep;126(3):e25-e27. doi: 10.1097/AOG.0000000000001049. PMID 26287789
- [Background] Wright D, Syngelaki A, Akolekar R, Poon LC, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal characteristics and medical history. Am J Obstet Gynecol. 2015 Jul;213(1):62.e1-62.e10. doi: 10.1016/j.ajog.2015.02.018. Epub 2015 Feb 25. PMID 25724400
- [Background] O'Gorman N, Wright D, Syngelaki A, Akolekar R, Wright A, Poon LC, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal factors and biomarkers at 11-13 weeks gestation. Am J Obstet Gynecol. 2016 Jan;214(1):103.e1-103.e12. doi: 10.1016/j.ajog.2015.08.034. Epub 2015 Aug 19. PMID 26297382
- [Background] O'Gorman N, Wright D, Poon LC, Rolnik DL, Syngelaki A, de Alvarado M, Carbone IF, Dutemeyer V, Fiolna M, Frick A, Karagiotis N, Mastrodima S, de Paco Matallana C, Papaioannou G, Pazos A, Plasencia W, Nicolaides KH. Multicenter screening for pre-eclampsia by maternal factors and biomarkers at 11-13 weeks' gestation: comparison with NICE guidelines and ACOG recommendations. Ultrasound Obstet Gynecol. 2017 Jun;49(6):756-760. doi: 10.1002/uog.17455. PMID 28295782
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Plasencia W, Maiz N, Poon L, Yu C, Nicolaides KH. Uterine artery Doppler at 11 + 0 to 13 + 6 weeks and 21 + 0 to 24 + 6 weeks in the prediction of pre-eclampsia. Ultrasound Obstet Gynecol. 2008 Aug;32(2):138-46. doi: 10.1002/uog.5402. PMID 18634131
- [Background] Poon LC, Zymeri NA, Zamprakou A, Syngelaki A, Nicolaides KH. Protocol for measurement of mean arterial pressure at 11-13 weeks' gestation. Fetal Diagn Ther. 2012;31(1):42-8. doi: 10.1159/000335366. Epub 2012 Jan 13. PMID 22248988
- [Derived] Chen Y, Nguyen-Hoang L, Dinh LT, Nguyen DA, Pooh RK, Shiozaki A, Zheng M, Hu Y, Ma R, Kusuma A, Wataganara T, Choolani MA, Kaneko M, Luewan S, Chang TY, Chaiyasit N, Nanthakomon T, Jiang Y, Shaw SW, Leung WC, Mohamad AS, Aguilar A, Lau SL, Lee NMW, Liu J, Sahota DS, Chong MKC, Papastefanou I, Poon LC. Effect of aspirin on small for gestational age neonates in pregnancies at high-risk for preeclampsia: a secondary analysis of a cluster randomised clinical trial. Lancet Reg Health West Pac. 2025 Jun 5;59:101582. doi: 10.1016/j.lanwpc.2025.101582. eCollection 2025 Jun. PMID 40529816
- [Derived] Nguyen-Hoang L, Dinh LT, Tai AST, Nguyen DA, Pooh RK, Shiozaki A, Zheng M, Hu Y, Li B, Kusuma A, Yapan P, Gosavi A, Kaneko M, Luewan S, Chang TY, Chaiyasit N, Nanthakomon T, Liu H, Shaw SW, Leung WC, Mahdy ZA, Aguilar A, Leung HHY, Lee NMW, Lau SL, Wah IYM, Lu X, Sahota DS, Chong MKC, Poon LC; FORECAST Collaborators. Implementation of First-Trimester Screening and Prevention of Preeclampsia: A Stepped Wedge Cluster-Randomized Trial in Asia. Circulation. 2024 Oct 15;150(16):1223-1235. doi: 10.1161/CIRCULATIONAHA.124.069907. Epub 2024 Jun 26. PMID 38923439